CLINICAL TRIAL: NCT02872935
Title: Randomized Double Control Study to Assess the Efficacy of Administering 1 ml of Glycopyrrolate With the Spinal Dose in Minimizing Nausea and Vomiting in Patients Undergoing Cesarean Section Under Spinal Anesthesia
Brief Title: Minimizing Nausea and Vomiting During Spinals for CS
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Kokila N Thenuwara (Other)
Responsible Party: Sponsor-Investigator, Kokila N Thenuwara, Clinical Associate Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201301793
Record Dates: First submitted 2016-08-05; First posted 2016-08-19 (Estimated); Results first posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-05

CONDITIONS: Nausea; Vomiting
MeSH Terms: conditions — Nausea; Vomiting | interventions — Glycopyrrolate; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (2):
- Placebo: Normal Saline (Placebo Comparator): 1ml of Normal Saline will be given intravenously with the administering of the spinal dose
  Interventions: Drug: Normal Saline
- Glycopyrrolate group (Experimental): 1ml of Glycopyrrolate ( .2mg /ml) will be given intravenously with the administering of the spinal dose
  Interventions: Drug: Glycopyrrolate

INTERVENTIONS:
Drug: Glycopyrrolate — .2mg of Glycopyrrolate will be given intravenously with the administration of the spinal dose
  Other Names: Robinul
  Arms: Glycopyrrolate group
Drug: Normal Saline — 1ml of normal saline will be given intravenously with the administration of the spinal dose
  Other Names: .9% saline
  Arms: Placebo: Normal Saline

SUMMARY:
In parturients undergoing Cesarean section under spinal anesthesia, co-loading of 1 liter of crystalloids, with placing the spinal, along with administering a phenylephrine infusion and glycopyrrolate, enables placing a spinal with minimal perioperative nausea and vomiting and good intra and post-operative pain relief.

DETAILED DESCRIPTION:
The hypothesis of this study is as follows: In parturients undergoing Cesarean section under spinal anesthesia, co-loading of 1 liter of crystalloids, with placing the spinal, along with administering a phenylephrine infusion and glycopyrrolate, enables placing a spinal with minimal perioperative nausea and vomiting and good intra and post-operative pain relief.

The study group will receive phenylephrine infusion [dilution 100micrograms /cc] Rate of infusion 50micrograms /hour, approximately 30ml/hour To be started immediately after the placement of the spinal anesthetic Patient will also be given .4mg [1cc of glycopyrrolate], with the starting of the infusion

The control group, will receive phenylephrine infusion [dilution 100micrograms /cc] Rate of infusion 50micrograms /hour, approximately 30ml/hour To be started immediately after the placement of the spinal anesthetic Patient will also be given a placebo [1cc of N saline], with the starting of the infusion

Following the administration of the study drug/placebo, the patient will be monitored for severity of nausea , vomiting and pain at 5 minutes intervals from placement of the spinal to delivery of the baby, and then at 15 minutes intervals from delivery of the baby till the end of the surgery ( the cesarean section)

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant
2. American Society of Anesthesiologists risk classification I and II
3. Age > 18 years
4. Non-laboring
5. Patients with elective cesarean sections

Exclusion Criteria:

1. Non- English speakers
2. Height < 4' 11"
3. BMI >40 Kg/ mm
4. Antiemetic drug use in the 24 hours prior to cesarean delivery,
5. Hypertensive diseases of pregnancy
6. Chronic hypertension receiving antihypertensive treatment
7. Any other physical or psychiatric condition that may impair their ability to cooperate with study data collection.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2015-05-15 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2016-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kokila N Thenuwara, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No
Do not plan to share data

REFERENCES:
- [Background] Carvalho B, Cohen SE, Lipman SS, Fuller A, Mathusamy AD, Macario A. Patient preferences for anesthesia outcomes associated with cesarean delivery. Anesth Analg. 2005 Oct;101(4):1182-1187. doi: 10.1213/01.ane.0000167774.36833.99. PMID 16192541
- [Background] Abouleish EI, Rashid S, Haque S, Giezentanner A, Joynton P, Chuang AZ. Ondansetron versus placebo for the control of nausea and vomiting during Caesarean section under spinal anaesthesia. Anaesthesia. 1999 May;54(5):479-82. doi: 10.1046/j.1365-2044.1999.00798.x. PMID 10995148
- [Background] Harmon D, Ryan M, Kelly A, Bowen M. Acupressure and prevention of nausea and vomiting during and after spinal anaesthesia for caesarean section. Br J Anaesth. 2000 Apr;84(4):463-7. doi: 10.1093/oxfordjournals.bja.a013471. PMID 10823097
- [Derived] Griffiths JD, Gyte GM, Popham PA, Williams K, Paranjothy S, Broughton HK, Brown HC, Thomas J. Interventions for preventing nausea and vomiting in women undergoing regional anaesthesia for caesarean section. Cochrane Database Syst Rev. 2021 May 18;5(5):CD007579. doi: 10.1002/14651858.CD007579.pub3. PMID 34002866

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo: Normal Saline | Glycopyrrolate Group
Started | 11 | 11
Completed | 11 | 10 (One subject consented but did no proceed with the study.)
Not Completed | 0 | 1
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo: Normal Saline | Glycopyrrolate Group | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 11 | 22
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Reported Nausea
Description: Did the subject report nausea? The subject will respond with yes or no.
Time Frame: From the administration of the spinal anesthesia to delivery of baby - Total time 90minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo: Normal Saline | Glycopyrrolate Group
Number analyzed (Participants) | 11 | 11
Participants | 8 | 7

2. Primary Outcome: Number of Participants Who Experienced Vomiting.
Description: This measure is observed by care team. Reported as vomiting, yes or no.
Time Frame: From the administration of the spinal anesthesia to delivery of baby; Total time 90minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo: Normal Saline | Glycopyrrolate Group
Number analyzed (Participants) | 11 | 11
Participants | 4 | 2

ADVERSE EVENTS:
Arm/Group | Placebo: Normal Saline | Glycopyrrolate Group
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes